CLINICAL TRIAL: NCT05230979
Title: Effect of Common Bean Baked Snack (Phaseolus Vulgaris L.) Consumption on Blood Lipid Levels and Hormones Regulating Appetite and Satiety: Randomized Crossover Clinical Trials
Brief Title: Evaluation of Common Bean Baked Snack Consumption on Subjective Satiety, Energy Intake and Glycemic Response in People With Overweight and Normal Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: Centro de Investigación y Asistencia en Tecnología y Diseño del Estado de Jalisco (Unknown)
Responsible Party: Principal Investigator, Alejandro Escobedo Avila, Principal Investigator, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CI-09620b
Record Dates: First submitted 2022-01-17; First posted 2022-02-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Overweight; Healthy
Keywords: Functional food; Common bean; Snack; Cooked beans
MeSH Terms: conditions — Overweight | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal weight (Experimental): People with normal weight will consume 40 g of common bean baked snack, cooked beans or white bread for a single occasion.
  Interventions: Other: Common bean baked snack; Other: Cooked beans; Other: White bread
- Overweight (Experimental): People with overweight will consume 40 g of common bean baked snack, cooked beans or white bread for a single occasion.
  Interventions: Other: Common bean baked snack; Other: Cooked beans; Other: White bread
- Glycemic index (Experimental): Determination of glycemic index under the ISO 26642:2010.
  Interventions: Other: Anhydrous glucose (first session) (for glycemic index determination); Other: Anhydrous glucose (second session) (for glycemic index determination); Other: Common bean baked snack (for glycemic index determination)

INTERVENTIONS:
Other: Common bean baked snack — Participants with normal weight (n=18) and with overweight (n=18) will attend the institute after 10-14 h fasting. Initially, they are going to complete a physical activity questionnaire, and the first visual analog scale (VAS) of subjective satiety questionnaire followed by a finger-prick blood sample. Immediately, they will be instructed to consume 40 g of the preload (common bean baked snack, cooked beans or white bread) along with 100 mL of water within 10 min. The VAS and blood glucose will be measured every 15 min after starting to eat the test food. Another VAS will be used to assess the palatability of the preload products. After 45 min, an ad libitum meal consisting of freshly prepared sandwiches and 250 mL of water will be served in a single portion. Finally, the VAS of subjective satiety is going to be assessed again.
  Arms: Normal weight; Overweight
Other: Cooked beans — Participants with normal weight (n=18) and with overweight (n=18) will attend the institute after 10-14 h fasting. Initially, they are going to complete a physical activity questionnaire, and the first visual analog scale (VAS) of subjective satiety questionnaire followed by a finger-prick blood sample. Immediately, they will be instructed to consume 40 g of the preload (common bean baked snack, cooked beans or white bread) along with 100 mL of water within 10 min. The VAS and blood glucose will be measured every 15 min after starting to eat the test food. Another VAS will be used to assess the palatability of the preload products. After 45 min, an ad libitum meal consisting of freshly prepared sandwiches and 250 mL of water will be served in a single portion. Finally, the VAS of subjective satiety is going to be assessed again.
  Arms: Normal weight; Overweight
Other: White bread — Participants with normal weight (n=18) and with overweight (n=18) will attend the institute after 10-14 h fasting. Initially, they are going to complete a physical activity questionnaire, and the first visual analog scale (VAS) of subjective satiety questionnaire followed by a finger-prick blood sample. Immediately, they will be instructed to consume 40 g of the preload (common bean baked snack, cooked beans or white bread) along with 100 mL of water within 10 min. The VAS and blood glucose will be measured every 15 min after starting to eat the test food. Another VAS will be used to assess the palatability of the preload products. After 45 min, an ad libitum meal consisting of freshly prepared sandwiches and 250 mL of water will be served in a single portion. Finally, the VAS of subjective satiety is going to be assessed again.
  Arms: Normal weight; Overweight
Other: Anhydrous glucose (first session) (for glycemic index determination) — Participants with normal weight or overweight (n=10) will attend the institute after 10-14 h fasting. At first, two baseline finger-prick blood samples will be collected with 5 min between the samples. Then, they are going to consume a reference glucose solution containing 25 g of anhydrous glucose per 250 mL of water within 12-15 min. Later, finger-prick blood samples will be taken at 15, 30, 45, 60, 90 and 120 min after starting to drink the reference glucose solution. Areas under the glucose response curves (iAUC) will be calculated using the trapezoidal rule, ignoring the areas below the fasting value.
  Arms: Glycemic index
Other: Anhydrous glucose (second session) (for glycemic index determination) — Participants with normal weight or overweight (n=10) will attend the institute after 10-14 h fasting. At first, two baseline finger-prick blood samples will be collected with 5 min between the samples. Then, they are going to consume 54 g of common bean baked snack with 250 mL of water within 12-15 min. Later, finger-prick blood samples will be taken at 15, 30, 45, 60, 90 and 120 min after starting to eat the test food. Areas under the glucose response curves (iAUC) will be calculated using the trapezoidal rule, ignoring the areas below the fasting value.
  Arms: Glycemic index
Other: Common bean baked snack (for glycemic index determination) — Participants with normal weight or overweight (n=10) will attend the institute after 10-14 h fasting. At first, two baseline finger-prick blood samples will be collected with 5 min between the samples. Then, they are going to consume 54 g of common bean baked snack with 250 mL of water within 12-15 min. Later, finger-prick blood samples will be taken at 15, 30, 45, 60, 90 and 120 min after starting to eat the test food. Areas under the glucose response curves (iAUC) will be calculated using the trapezoidal rule, ignoring the areas below the fasting value.
  Arms: Glycemic index

SUMMARY:
Introduction: Overweight and obesity are associated with an unbalanced energy intake caused by unhealthy dietary habits, including a constant consumption of energy-dense foods, saturated and trans fats, refined sugars, along with a deficient protein and dietary fiber intake. Pulse consumption has been demonstrated to improve long-term body weight management. Despite these benefits, in several regions, the consumption of pulses does not meet the local recommendations. Consequently, pulse research has increased widely in order to provide food alternatives reformulated with pulses to promote their consumption.

Hypothesis: The consumption of a common bean baked snack (Phaseolus vulgaris L.) and cooked beans increases satiety, reduces energy intake and produce a low glycemic response in people with overweight and normal weight.

Objectives: Evaluate the acute effect of a common bean baked snack and cooked bean consumption on subjective satiety and energy intake in people with overweight and normal weight.

Material and Methods: Randomized crossover clinical trial, 18 subjects with normal weight and 18 subjects with overweight, 18-50 years old, consumption of 40 g of common bean baked snack, cooked beans and white bread (control). Subjective satiety, energy intake and glycemic response.

* Intervention A: Common bean baked snack.
* Intervention B: Cooked beans.
* Control: White bread.

Additionally, the glycemic index will be determined under the International Organization for Standardization (ISO) 26642:2010.

10 subjects with normal weight or overweight, 18-50 years old, consumption of 54 g of common bean baked snack and 25 g of anhydrous glucose.

* Intervention A: Common bean baked snack.
* Control: Anhydrous glucose

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 29.9 kg/m2,

Exclusion Criteria:

* Pregnancy,
* Lactation,
* Established plans to lose or gain weight in the next three weeks,
* Surgical event or modification of diet or physical activity in the last three months,
* Diagnosis of diabetes, cancer, cardiovascular disease, gastrointestinal disorder, pancreatitis, kidney, liver or thyroid disease,
* Eating disorder,
* Smoking or drug use,
* Sensitivity for common bean consumption,
* Pharmacological treatment or consumption of non-prescription drugs, herbal or nutritional supplements known to modify appetite or satiety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Satiety | 45 minutes period, every 15 min after ingestion of the test meal.
  Subjective satiety will be measured using a 100-mm visual analogue scale [0 mm (not at all) - 100 mm (completely)] at 0, 15, 30 and 45 minutes after ingestion of the test meals. The scale comprises different perceptions of satiety including: hunger, fullness, prospective food intake, and thirst.
Ad libitum energy intake (kcal) | 45 minutes after ingestion of the test meal.
  Participants will consume sandwiches until they feel comfortably satisfied. The calories consumed will be calculated from the difference in weight of the initial and final portions of the sandwiches, using the nutritional information on the label of the package of each ingredient.
0-45 minutes Glycemic response | 0, 15, 30 and 45 minutes after ingestion of the test meal.
  Capillary blood glucose (mg/dL)
0-120 minutes Glycemic response | 0, 15, 30, 45, 60, 90, 120 minutes after ingestion of the test meal.
  Capillary blood glucose (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar A. Rivera León, PhD, Principal Investigator — Departamento de Biología Molecular y Genómica, Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara
Locations (1):
- Departamento de Biología Molecular y Genómica, Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Non-shareable data.